CLINICAL TRIAL: NCT04504500
Title: Reducing the Cesarean Section Rates and Enhancing Vaginal Delivery in Greece Through Educational, Behavioral and Organizational Interventions in Labor Management: a Stepped-Wedge Randomized Controlled Trial (ENGAGE Trial)
Brief Title: Reducing Cesarean Section Rates and Enhancing Vaginal Delivery in Greece: a Stepped-Wedge Randomized Controlled Trial
Acronym: ENGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Society of Obstetrics and Gynecology (Other)
Collaborators: St George's, University of London (Other); A. G. Leventis Foundation (Unknown); National and Kapodistrian University of Athens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 129/29062018
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Cesarean Section Rates
Keywords: cesarean section; vaginal delivery; birth; Greece; maternal morbidity; perinatal morbidity; ENGAGE trial; stepped-wedge trial; intervention; guideline
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: The trial herein discussed is a stepped-wedge cluster randomized trial involving random and sequential crossover of maternity units (clusters) from observation (routine practice, control) to intervention (educational, behavioral and organizational interventions), until all maternity units (clusters) have been exposed. The primary and secondary outcomes of the two phases (observation and intervention) are compared.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation phase (No Intervention): Routine practice assessment
- Intervention phase (Active Comparator): Clinical practice assessment after the application of the trial's educational, behavioral and organizational interventions
  Interventions: Behavioral: HSOG guidelines application; Behavioral: Interactive workshops and courses; Behavioral: Feedback through follow-up meetings; Behavioral: Robson criteria usage; Behavioral: Access to live real-time statistics; Behavioral: Attendance of local cesarean section meetings; Behavioral: Attendance of local CTG interpretation meetings; Behavioral: Reminders of proper clinical practice; Other: HSOG guidelines implementation; Other: Interactive workshops and courses training; Other: Implementation of Robson criteria classification; Other: Live real-time statistics online platform; Other: Local cesarean section meetings; Other: Local CTG interpretation meetings; Other: Follow-up meetings

INTERVENTIONS:
Behavioral: HSOG guidelines application — In their practice, as regards the mode of delivery, obstetricians are encouraged to conform to the three guidelines and two consent forms published by the Hellenic Society of Obstetrics and Gynecology (HSOG). The members of the appointed Steering Committee and/or local opinion leaders will discuss and disseminate these guidelines among the professional staff in the respective maternity units, providing them with the opportunity to identify specific barriers, overcome them, and develop an implementation timetable.
  Arms: Intervention phase
Behavioral: Interactive workshops and courses — The workshops and courses will give instruction in indications for cesarean section and clinical scenarios, physiology-based cardiotocography (CTG) interpretation, obstetric emergencies (with topics including breech delivery, trial of labor after cesarean, delivery of twins, induction and augmentation of labor), organization of the labor ward, as well as launching of regular cesarean section and CTG meetings with review of the patient notes. The workshops will last four days and will be conducted by experienced trainers. The expectation is that the obstetricians will gain very considerable knowledge and skills, which will enable them to subsequently follow these practices safely and competently.
  Arms: Intervention phase
Behavioral: Feedback through follow-up meetings — Regular follow-up meetings with members of the steering committee and local opinion leaders throughout the intervention period will enhance compliance with the guidelines. Feedback with positive phrasing will be incorporated to meet local needs.
  Arms: Intervention phase
Behavioral: Robson criteria usage — Obstetricians are set to a routine to enable them to use the Robson 10-group classification criteria for cesarean sections and obtain feedback on the unit's cesarean section rates monthly. They thus know which category is higher and can be reduced further.
  Arms: Intervention phase
Behavioral: Access to live real-time statistics — Live real-time statistics provided by an online platform, on a regular basis, is expected to improve adherence, through regular feedback. Each unit will see other units' statistics by means of an anonymous reporting system. This repetition will create silent signals that will remind the participating obstetricians to remain on task.
  Arms: Intervention phase
Behavioral: Attendance of local cesarean section meetings — Local cesarean section meetings will be held weekly, in each unit. The members of the steering committee or local opinion leaders may actively participate in these meetings. Local obstetricians learn to judiciously adapt standard medical practices, thereby avoiding unnecessary medical interventions. This is a way to further enhance compliance, as during the discussions the behavior expected of the obstetricians is clearly stated by the participating opinion leaders.
  Arms: Intervention phase
Behavioral: Attendance of local CTG interpretation meetings — Local CTG interpretation meetings will be held weekly, in each unit, during which all "abnormal" CTG cases that led to cesarean section will be reviewed and discussed. Members of the Steering Committee or local opinion leaders may actively participate in these meetings. Obstetricians are encouraged to reflect on their medical practice through judicious physiology-based CTG interpretation.
  Arms: Intervention phase
Behavioral: Reminders of proper clinical practice — Effective and reliable reminders concerning optimal obstetric practice will be placed in labor wards, staff rooms, patient notes, vaginal birth packages and above theater hand washers. There will be short messages with positive phrasing regarding the benefits of vaginal birth, thus reminding birth attendants to reduce unnecessary cesarean sections. Relevant SMS (short message service) will be sent to the participating obstetricians' mobiles on a regular basis, so as to motivate them via non-verbal signals.
  Arms: Intervention phase
Other: HSOG guidelines implementation — There will be application in daily practice of three guidelines and two consent forms pertaining to the mode of delivery published by HSOG. Obstetricians are informed on evidence-based medicine in obstetrics and provided with a structured and safe approach to labor management. The members of the appointed Steering Committee and/or local opinion leaders discuss and disseminate the guidelines among the professional staff at the respective maternity units, answer questions, and make available their knowledge and experience. Adoption of guidelines by the participating unit helps to establish clear, consistent rules that are direct and simple, and obstetricians are asked to embrace fully justified medical practice.
  Other Names: Educational and organizational intervention
  Arms: Intervention phase
Other: Interactive workshops and courses training — The workshops and courses will provide instruction in indications for cesarean section and case scenarios, physiology-based CTG interpretation, obstetric emergencies (with topics including breech delivery, trial of labor after cesarean, delivery of twins, induction and augmentation of labor), organization of labor ward and launching of cesarean section and CTG meetings. This type of formal training provides problem-solving strategies, using mnemonics, that are critical in emergencies and that also aid in learning and retaining the skills being taught. Functional and social skills that directly affect decision-making and effectiveness are addressed. Thus, units adopt a continuous educational procedure for their staff, enhancing their confidence when dealing with labor emergencies and redesigning labor management plans, so as to ensure high-level obstetric services.
  Other Names: Educational and organizational intervention
  Arms: Intervention phase
Other: Implementation of Robson criteria classification — Use will be implemented of an online application embedded in the REDCap electronic database questionnaire with Robson 10-group classification criteria and feedback on the unit's cesarean section rates monthly, so as to know which category is higher and can be reduced further. This change in the unit's practice will introduce a new medical reporting and audit system that can detect unjustified medical procedures much more easily.
  Other Names: Educational and organizational intervention
  Arms: Intervention phase
Other: Live real-time statistics online platform — Live real-time statistics provided on a regular basis by an online platform will provide feedback and essential information. Each unit will see other units' statistics using an anonymous reporting system. This information can trigger self-generative learning strategies and help obstetricians to become more effective learners.
  Other Names: Educational intervention
  Arms: Intervention phase
Other: Local cesarean section meetings — Local cesarean section meetings will be held weekly in each unit. The members of the Steering Committee or local opinion leaders may actively participate in these meetings. The unit's staff can hear about both justified and unnecessary surgical procedures and draw informed conclusions as to the optimal procedure in similar cases. They will also have the opportunity to actively participate in an elaborative problem-solving discussion. These meetings when routinely conducted, provide feedback and audit resources to help improve performance and further enhance compliance.
  Other Names: Educational and organizational intervention
  Arms: Intervention phase
Other: Local CTG interpretation meetings — Local CTG interpretation meetings will be held weekly, in each unit during which all "abnormal" CTG cases that led to cesarean section will be reviewed and discussed. Members of the Steering Committee or local opinion leaders may actively participate in these meetings offering coaching and counseling services in decision-making. Through elaborative discussion the staff will improve their knowledge and skills in correct CTG interpretation, thus preventing unnecessary interventions, such as cesarean sections.
  Other Names: Educational and organizational intervention
  Arms: Intervention phase
Other: Follow-up meetings — Regular follow-up meetings of the participating obstetricians with members of the steering committee and local opinion leaders throughout the intervention period will enhance compliance with the guidelines. Establishment of commonly accepted practice augments the homogeneity of clinical action plans and team work in the unit.
  Other Names: Organizational intervention
  Arms: Intervention phase

SUMMARY:
It is becoming increasingly apparent that there is an urgent need to systematically investigate the rising cesarean section (CS) rates in Greece and develop interventions to substantially reduce these rates. In this trial, to be conducted in Greece, the obstetricians will be exposed to educational, behavioral and/or organizational interventions while managing labor. The trial is expected to yield new information about effective interventions to reduce unnecessary cesarean sections in Greece, hopefully leading the way to their reduction worldwide.

DETAILED DESCRIPTION:
The present study explains the planned implementation of a stepped-wedge trial in Greek maternity units. Twenty-two maternity units in Greece will participate in the trial involving 20,000 to 25,000 births, with two of the units entering the intervention period each month (stepped randomization). The maternity units will apply the interventions for a period of 6-16 months, depending on the time they enter the intervention stage of the trial. There will also be an initial baseline phase of the trial, lasting from 3 to 13 months; this phase will include observation and data collection of routine obstetric practices. The interventions are based on educational, behavioral and organizational modifications and will include the implementation of the Hellenic Society of Obstetrics and Gynecology (HSOG) guidelines on labor management and targeted training in cardiotocography (CTG), obstetric emergencies, and the classification of cesarean section through Robson criteria. During the trial period, the rates and indications for cesarean sections will be available to participating units on a live platform, using an anonymous reporting system. Participating obstetricians will be able to see their own and other units' performance and also get feedback on their rates. Τhe final three-month phase of the trial will be devoted to completion of questionnaires by the participating obstetricians. The total estimated duration of the trial will be 22 months. The primary outcome assessed will be the change in cesarean section rate and the secondary outcomes will be maternal and neonatal morbidity and mortality. The intervention and control periods will be compared using mixed effects logistic regression with adjustment for any underlying secular trends.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 5 years' provision of obstetric services for the participating units.
* Top 22 units in Greece according to the number of deliveries and the type of unit (National Health System, private, university) and the unit's willingness to participate.
* Up to 11 obstetricians in each unit (based on the number of deliveries and their willingness to participate)
* Consent obtained from all participating professionals
* Consent obtained from all participating women

Exclusion Criteria:

* None

Ages: 14 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 6029 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Cesarean section rate | Admission to maternity unit to time of vaginal or cesarean birth
  Number of cesarean section deliveries in the study period divided by the number of live vaginal and cesarean births

SECONDARY OUTCOMES:
Maternal morbidity | During labor and 40 days to 3 months after delivery
  Incidence of maternal complications in labor and postpartum
Perinatal and neonatal morbidity | During labor and 40 days to 3 months after delivery
  Incidence of perinatal and neonatal complications in labor and postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Vrachnis, Prof Ob/Gyn, Principal Investigator — Hellenic Society of Obstetrics and Gynecology
Locations (1):
- All participating units, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
Study data may be shared upon chief investigator's decision after reasonable request and up to 8 year after the conclusion of the trial.

REFERENCES:
- [Background] Vrachnis N, Vlachadis N, Iliodromiti Z, Vlachadi M, Creatsas G. Greece's birth rates and the economic crisis. Lancet. 2014 Feb 22;383(9918):692-3. doi: 10.1016/S0140-6736(14)60252-X. No abstract available. PMID 24560050
- [Background] Betran AP, Torloni MR, Zhang JJ, Gulmezoglu AM; WHO Working Group on Caesarean Section. WHO Statement on Caesarean Section Rates. BJOG. 2016 Apr;123(5):667-70. doi: 10.1111/1471-0528.13526. Epub 2015 Jul 22. No abstract available. PMID 26681211
- [Background] Vlachadis N, Vrachnis N, Economou E. Fertility treatments and multiple births in the United States. N Engl J Med. 2014 Mar 13;370(11):1069-70. doi: 10.1056/NEJMc1400242. No abstract available. PMID 24620878
- [Background] Betran AP, Ye J, Moller AB, Zhang J, Gulmezoglu AM, Torloni MR. The Increasing Trend in Caesarean Section Rates: Global, Regional and National Estimates: 1990-2014. PLoS One. 2016 Feb 5;11(2):e0148343. doi: 10.1371/journal.pone.0148343. eCollection 2016. PMID 26849801
- [Background] Vlachadis N, Iliodromiti Z, Creatsas G, Vrachnis N. Preterm birth time trends in Europe: the worrying case of Greece. BJOG. 2014 Feb;121(3):372-3. doi: 10.1111/1471-0528.12529. No abstract available. PMID 24428453
- [Background] The Lancet. Stemming the global caesarean section epidemic. Lancet. 2018 Oct 13;392(10155):1279. doi: 10.1016/S0140-6736(18)32394-8. No abstract available. PMID 30322560
- [Background] Vrachnis N, Iliodromiti S, Samoli E, Iliodromiti Z, Dendrinos S, Creatsas G. Maternal mortality in Greece, 1996-2006. Int J Gynaecol Obstet. 2011 Oct;115(1):16-9. doi: 10.1016/j.ijgo.2011.04.014. Epub 2011 Jul 23. PMID 21788018
- [Background] Chen I, Opiyo N, Tavender E, Mortazhejri S, Rader T, Petkovic J, Yogasingam S, Taljaard M, Agarwal S, Laopaiboon M, Wasiak J, Khunpradit S, Lumbiganon P, Gruen RL, Betran AP. Non-clinical interventions for reducing unnecessary caesarean section. Cochrane Database Syst Rev. 2018 Sep 28;9(9):CD005528. doi: 10.1002/14651858.CD005528.pub3. PMID 30264405
- [Background] Vrachnis N, Vlachadis N. Maternal mortality estimates. Lancet. 2014 Dec 20;384(9961):2210. doi: 10.1016/S0140-6736(14)62423-5. Epub 2014 Dec 19. No abstract available. PMID 25625395
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Background] Vlachadis N, Vrachnis N, Tsikouras P, Mastorakos G, Iliodromiti Z. Birth rates by maternal age in Greece: background, trends and future perspectives. J Reprod Med. 2015 Mar-Apr;60(3-4):183-4. No abstract available. PMID 25898486
- [Derived] Vrachnis N, Antonakopoulos N, von Dadelszen P, Vidler M, Maroudias G, Bone J, Sandhu A, Loukas N, Magee L, Roussos N, Kassaris S, Fotiou A, Zygouris D, Adonakis G, Akrivis C, Antsaklis A, Athanasiadis A, Bontis N, Daniilidis A, Daponte A, Daskalakis G, Deligeoroglou E, Dinas K, Drakakis P, Gerede A, Grimbizis G, Iacovidou N, Kambas N, Katasos T, Katsetos C, Katsikis I, Makrigiannakis A, Matalliotakis M, Messini C, Mikos T, Nikolettos N, Pados G, Paschopoulos M, Patsouras K, Siahanidou S, Sioulas V, Skentou C, Stavros S, Temmerman M, Tsikouras P, Tsitsis V, Vlahos N, Rodolakis A, Papageorghiou A, Loutradis D. ENhancinG vAGinal dElivery in Greece through educational and behavioral interventions among maternity care providers regarding labor management: the ENGAGE stepped-wedge randomized prospective trial protocol. Trials. 2024 Aug 19;25(1):548. doi: 10.1186/s13063-024-08263-x. PMID 39155367
- See also: Trial webpage — https://emgetrial.gr/